CLINICAL TRIAL: NCT02928354
Title: A Randomized Open Label Three-Way Crossover Study in Healthy Male Volunteers to Investigate the Effect of Particle Size on Pharmacokinetics Following a Single Inhaled Dose of AZD7594 Via a Dry Powder Inhaler
Brief Title: A Study to Assess the Effect of Particle Size of AZD7594 on Pharmacokinetics (PK) After a Single Inhaled Dose When Administered Using the Dry Powder Inhaler in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3741C00006
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Asthma, Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Asthma; Chronic obstructive pulmonary disease (COPD); Healthy volunteers; Pharmacokinetics (PK); Bioavailability; AZD7594; Safety; Tolerability
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A - AZD7594 (Experimental): Treatment A - AZD7594 inhalation powder Particle size Large
  Interventions: Drug: Treatment A - AZD7594
- Treatment B - AZD7594 (Experimental): Treatment B - AZD7594 inhalation powder Particle size Medium
  Interventions: Drug: Treatment B - AZD7594
- Treatment C - AZD7594 (Experimental): Treatment C - AZD7594 inhalation powder Particle size Small
  Interventions: Drug: Treatment C - AZD7594

INTERVENTIONS:
Drug: Treatment A - AZD7594 — Particle size Large as a single inhaled dose of 440 µg (nominal dose), administered via DPI
  Arms: Treatment A - AZD7594
Drug: Treatment B - AZD7594 — Particle size Medium as a single inhaled dose of 440 µg (nominal dose), administered via DPI
  Arms: Treatment B - AZD7594
Drug: Treatment C - AZD7594 — Particle size Small as a single inhaled dose of 440 µg (nominal dose), administered via DPI
  Arms: Treatment C - AZD7594

SUMMARY:
This study is an open label, randomized, three-way crossover study to assess the effect of particle size on the PK and safety of single inhaled doses of AZD7594 in healthy subjects (males aged 18 to 55 years [inclusive]). The study will be performed at a single study center.

DETAILED DESCRIPTION:
The study will comprise:

* A Screening period of maximum 28 days.
* Three treatment periods during which subjects will be resident prior to the evening meal the 1 day before dosing with AZD7594 (Day -1) until at least 48 hours after dosing; discharged on the morning of Day 3. Subjects will then return for ambulatory visits 72, 96, 144 and 240 hours after dosing, (Day 4, Day 5, Day 7 and Day 11 respectively).
* A final Follow-up Visit within 10 days after the last administration of AZD7594. This visit will coincide with the last PK sample collection on Day 11 after the last Treatment Period.

There will be a minimum wash-out period of 21 and maximum of 28 days between each dose administration.

Subjects will attend a Screening Visit within 28 days before receiving their first dose of AZD7594, if they are found to be eligible, they return for Treatment Period 1, when they will have baseline assessments, and then will be randomized into one of the 6 treatments sequences. For each Treatment Period, the subjects will receive their investigational medicinal product (IMP) dose in the morning of Day 1, will have further assessments for 48 hours after dosing (residential period) and will return to the study center for ambulatory visits 72, 96, 144 and 240 hours after dosing, (Day 4, Day 5, Day 7 and Day 11 respectively).

Each subject will receive AZD7594 as a single inhaled dose of 440 µg (nominal dose) of each of the following treatments, administered via Dry powder inhaler (DPI):

* Treatment A: Particle size Large
* Treatment B: Particle size Medium
* Treatment C: Particle size Small Each subject will be involved in the study for up to 12 weeks (up to 4 weeks for enrollment and 8 weeks of active study and Follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Subjects should be willing to follow reproductive restrictions to prevent pregnancy and drug exposure of a female partner and refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of IMP.
5. Be able to inhale from the DPI devices according to given instructions.
6. Subjects must read, speak and understand German language.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
4. Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results, at screening and first admission to the study unit as judged by the PI.
5. Any clinically significant abnormal findings in vital signs at screening and first admission to the study unit, as judged by the PI. Abnormal vital signs, after 10 minutes supine rest, defined as any of the following: - Systolic BP (SBP) < 90 mmHg or > 140 mmHg - Diastolic BP (DBP) < 50 mmHg or > 90 mmHg - Heart rate < 45 or > 90 beats per minute.
6. Any clinically significant abnormalities on 12-lead ECG at screening and first admission to the study unit, as judged by the PI.
7. Any positive result on screening for serum hepatitis surface antigen or antiHBc antibody suggestive of hepatitis B infection, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
8. Known or suspected history of drug abuse, as judged by the PI.
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7594.
12. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
13. Subjects who are not able to perform correct spirometry tests at screening.
14. Subjects with forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) <80% predicted (calculated) values and FEV1/FVC ratio <0.7 in pulmonary function test (spirometry) at Screening Visit.
15. Positive screen for drugs of abuse or cotinine at screening or on each admission to the study center or positive screen for alcohol on each admission to the study center.
16. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
17. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
18. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.
19. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
20. Subjects who have previously received AZD7594.
21. Judgment by the PI that the volunteer should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
22. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) | Pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of AUC in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC last) | Pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of AUC last in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Maximum observed plasma concentration (Cmax) | Pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of Cmax in healthy male volunteers after the administration of single inhaled dose of AZD7594.

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (tmax) | Pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of tmax in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t ½,λz) | Pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of t ½,λz in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Mean residence time from zero to infinity (MRT) | pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of MRT in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Terminal elimination rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) | Pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of λz in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Apparent total body clearance of drug from plasma after extravascular administration, estimated as dose divided by AUC (CL/F) | pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of CL/F in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Apparent volume of distribution during the terminal phase after extravascular administration estimated by dividing CL/F by λz (Vz/F) | pre-dose and at 15, 30, and 45 minutes, and 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48, 72, 96, 144 and 240 hours post dose
  Assessment of (Vz/F) in healthy male volunteers after the administration of single inhaled dose of AZD7594.
Adverse events (AEs) | Throughout the study ie. from screening (Day -28) upto follow up visit i.e.. 10 days after last IMP administration
  Assessment of the safety in terms of the incidences of the AEs after the administration of single inhaled dose of AZD7594.
Physical examination | On screening (Day -28), Day 1 to 3 and follow up visit i.e., 10 days after last IMP administration
  Assessment of the safety in terms of the physical examination after the administration of single inhaled dose of AZD7594.
Electrocardiogram (ECG) | Safety ECG will be performed prior to IMP administration and 1, 4 and 24 hours post-IMP administration on Day 1 of each Treatment Period
  Assessment of the safety in terms of the ECG after the administration of single inhaled dose of AZD7594.
Vital signs (systolic and diastolic blood pressure [BP], pulse rate) | Vital signs: pulse, blood pressure and oral body temperature will be measured, pre-dose and 1, 4, 24 hours post dose of each Treatment Period
  Assessment of the safety in terms of the Vital signs (systolic and diastolic blood pressure, pulse rate) after the administration of single inhaled dose of AZD7594.
Spirometry | On Day 1 of each Treatment Period spirometry will be performed pre-dose and at 0.5 and 1 hours post dose
  Assessment of the safety in terms of the spirometry after the administration of single inhaled dose of AZD7594.
Clinical laboratory assessments (hematology, clinical chemistry (including serum potassium and glucose) | Safety laboratory tests will be performed at screening, Day 1, Day 11, 240 h post dose and follow up visit
  Assessment of the safety in terms of the Clinical laboratory assessments (hematology, clinical chemistry (including serum potassium and glucose) after the administration of single inhaled dose of AZD7594.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas Körnicke, Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany